CLINICAL TRIAL: NCT05521776
Title: Impact of First-trimester Preeclampsia Screening on Perinatal and Maternal Morbidity : a Multicenter Randomized Trial
Brief Title: Impact of First-trimester Preeclampsia Screening on Perinatal and Maternal Morbidity (RANSPRE)
Acronym: RANSPRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other); INSERM, Epopé team (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: APHP211047; 2022-A00374-39 (Other: ID-RCB Number)
Record Dates: First submitted 2022-07-07; First posted 2022-08-30 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Preeclampsia (PE)
Keywords: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- With first trimester preeclampsia screening (Experimental): Risk assessment of developing preeclampsia between 11 and 14 WG based on maternal parameters, blood pressure measurement, Doppler measurements of the uterine arteries and maternal PlGF concentration. Patients at high risk of preeclampsia are treated with aspirin.
  Interventions: Procedure: First-trimester preeclampsia screening (FMF triple test)
- Without first trimester preeclampsia screening (No Intervention): Usual prenatal care

INTERVENTIONS:
Procedure: First-trimester preeclampsia screening (FMF triple test) — An algorithm assessing the risk of developing preeclampsia combining maternal parameters, blood pressure measurement, Doppler measurements of the uterine arteries and maternal PlGF concentrations.
  For women in the screening group, a Doppler study of the uterine arteries and a blood test to quantify PlGF concentrations will be performed within 2 days of randomization, allowing the risk to be calculated according to the screening test. For women with a positive screening test (i.e. predicted risk> 1/100), a treatment with aspirin will be prescribed at 160 mg/day, started as soon as possible and before 15 WG, and taken up to 36 WG, in the absence of contraindications. For women with negative screening, usual pregnancy monitoring without aspirin will be offered.
  Arms: With first trimester preeclampsia screening

SUMMARY:
The purpose of this study is to determine whether first-trimester screening for preeclampsia based on the FMF algorithm (a combination of maternal clinical, sonographic and biochemical parameters), improves maternal or perinatal health.

DETAILED DESCRIPTION:
Preeclampsia (PE) complicates 2% of pregnancies and is a leading cause of severe maternal and perinatal complications. There is no curative treatment, and the only recognized beneficial primary prevention is low-dose aspirin. Meta-analyses of randomized trials show that the administration of aspirin, started before 16 weeks of gestation (WG) and at the dosage of 100-160 mg/d in pregnant women at high risk of PE, is associated with a 50% to 60% reduction in the rates of PE, prematurity and perinatal mortality. The group of patients benefiting most from aspirin is pregnant women with a history of PE. That is why all guidelines recommend early preventive administration of aspirin in pregnant women with PE in a previous pregnancy. However, patients with a history of PE represent a small fraction of pregnant women, and PE mostly occurs in women who do not have a history of PE, especially nulliparas. Recently, several national societies decided to broaden the indications for aspirin prevention on the basis of the number of known maternal risk factors. These recommendations lead to a wide use of low-dose aspirin in up to 30% of pregnant women. In order to better target patients at risk of PE among all pregnant women, screening tests have been developed integrating clinical characteristics, uterine Doppler (UD) parameters and biomarkers in a single score. The study by Poon et al. paved the way for early detection of PE. An algorithm based on maternal characteristics, UD parameters and serum levels of PlGF and PAPP-A between 11 and 14 WG yielded detection rates of 93% and 36% for the prediction of early- and late-onset PE, respectively, at 5% false-positive rate (FPR), which were superior to the detection rates of the traditional checklist-based approach, which relies on maternal factors only. This algorithm developed by the Fetal Medicine Foundation (FMF) has since evolved and is now integrated in the combined test for PE screening known as the FMF triple test (a combination of maternal characteristics with mean arterial pressure (MAP), uterine artery pulsatility index (UtA-PI), and serum PlGF). In a subsequent study using a risk cutoff of 1 in 100 for the predicted probability of preterm PE, a screen-positive rate of 10% has been reported, with detection rates for early-onset, preterm, and term PE of 88%, 69%, and 40%, respectively.

Recently, the ASPRE study evaluated the impact of aspirin in patients identified at high risk of PE on the basis of this FMF test. Screening was offered to 26,941 women and identified 2,641 high-risk patients of whom 1,776 were randomized to aspirin or placebo. This trial showed a reduction in the incidence of PE <37 WG, occurring in 13/798 in the aspirin group versus 35/822 in the placebo group (p=0.004), but with no significant effect on the overall rate of PE and most importantly on perinatal morbidity. Screening had to be applied to almost 27,000 women for a benefit of 22 avoided cases of preterm PE, with no demonstrated effect on the health of the women and children. The ASPRE study is important but does not demonstrate the benefit of routinely implementing PE screening in the general population. Indeed, there is currently no randomized study comparing a group of women to which the screening procedure would be applied to a group of women without screening, the only design able to provide strong evidence of a benefit. In addition, implementing a national screening program in pregnant women may induce adverse events, especially iatrogenicity (more hospitalizations, more ultrasound examinations, more consultations) and anxiety. Such a screening program is also associated with an increase of direct and indirect health costs.

To consider implementing screening for PE in the general population, it is then essential to demonstrate its benefits on robust health outcomes and not only on the PE diagnosis, as well as to assess its potential adverse consequences and costs. This evaluation is all the more crucial since it is currently offered to an increasing number of women.

The RANSPRE study will therefore be the first trial to test the impact on perinatal and maternal health outcomes of first-trimester screening for preeclampsia associated with aspirin treatment of pregnant women screened at risk. A medical and economic evaluation allowing a cost-effectiveness analysis will also be carried out. The results of this study will constitute essential information relevant to the health care system that will guide policymaking for the prevention of PE in the general population of pregnant women.

The primary objective of the study is to evaluate the impact of first-trimester PE screening (FTPS) on the incidence of severe perinatal morbidity. The primary outcome will be severe perinatal morbidity defined by a composite criterion including at least one of the following: perinatal mortality (stillbirth at or after 20 WG or neonatal death within 7 days of life) or prematurity <34 WG or birth weight <3° percentile for gestational age.

Secondary objectives are: (i) to evaluate the impact of first-trimester PE screening on: the incidence of preeclampsia, the incidence of components of moderate and severe maternal morbidity, the incidence of components of moderate and severe perinatal morbidity; (ii) to evaluate the impact of first-trimester PE screening on potential adverse events: iatrogenicity, over-medicalization, women's satisfaction and anxiety status; (iii) to evaluate the economic impact of first-trimester PE screening on costs.

Patients will be recruited in 22 maternity centers at university hospitals in France. The inclusion period during pregnancy is between 11 WG and 14 WG. Eligible women will be identified in early pregnancy at their first prenatal visit in the maternity hospital, before or at the time of the first-trimester ultrasound. The FMF algorithm used in the study for PE screening is based on a combination of maternal clinical parameters (medical history, maternal characteristics, pregnancy characteristics, mean arterial pressure), sonographic parameters (uterine Doppler with measurement of mean pulsatility index) and biochemical parameters (PlGF concentration). Women agreeing to participate in the RANSPRE trial will be randomized either to the experimental group with first-trimester screening for PE or to the control group with usual care without screening for PE.

All patients will be asked to complete self-administered questionnaires at 20 (+/2) WG and during the postpartum period (within 30 days after delivery) assessing women's satisfaction and women's anxiety. These questionnaires will be collected for women included until 31/01/2025.. A notebook will be given to patients screened at risk and with aspirin prescription to monitor aspirin observance and to record potential side-effects related to aspirin.

An intention-to-treat analysis will be performed as the principal analysis.

ELIGIBILITY:
Inclusion Criteria :

* Pregnancy between 11 and 14 WG
* Age ≥18 years
* Affiliated to or beneficiary of a health insurance system (including AME)
* Signed informed consent

Exclusion Criteria :

* Gestational age <11 WG and >14 WG
* Known ectopic pregnancy
* Known non-ongoing pregnancy
* Known multiple pregnancy
* History of PE in a previous pregnancy
* Pregnancies complicated by major fetal abnormality identified at the first-trimester ultrasound if performed before randomization
* Absence of health insurance
* Contra-indication to aspirin (bleeding disorders such as von Willebrand's disease, active peptic ulceration, hypersensitivity to aspirin, active peptic ulceration, NSAID-exacerbated respiratory disease, severe liver or heart dysfunction)
* Women taking low-dose aspirin regularly before pregnancy (except ART indication)
* Age <18 years
* Poor understanding of the French language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14500 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-03-06 (Estimated)

PRIMARY OUTCOMES:
Severe perinatal morbidity | From birth up to 7 days of life
  The primary outcome is a composite criterion characterizing severe perinatal morbidity including one of the following criteria:
  * perinatal mortality: death of a fetus at or after 20 WG or weighing more than 500 g, or death of a newborn within the first 7 days of life.
  * prematurity < 34 WG: birth before 34 WG
  * birth weight < 3° percentile

SECONDARY OUTCOMES:
Incidence of preeclampsia | From inclusion up to discharge from hospital after delivery (max 30 days)
  PE defined as gestational hypertension (GH: systolic BP ≥140 and/or diastolic BP ≥90 mm Hg) and proteinuria ≥ 0.30 g/day (or PCr ratio ≥30 mg/mmol, or at least ++ on dipstick analysis if no 24-hour collection is available), at or after 20 WG and up to discharge from hospital after delivery. PE also defined according to the 2018 ISSHP in the absence of proteinuria in case of GH with maternal organ dysfunction: • creatinine ≥90 µmol/L • transaminases >40 IU/L • eclampsia, altered mental status, blindness, stroke, severe headache unresponsive to medication, and persistent visual scotomata) • platelet count <150000/μL, DIVC, hemolysis • Fetal weight <3° centile, abnormal umbilical artery Doppler (PI>90° centile), or stillbirth - Early-onset PE <34 WG, late-onset PE ≥34 WG - Superimposed pre-eclampsia when a woman with chronic hypertension develops proteinuria (in the absence of preexisting proteinuria) or any of the maternal organ dysfunction consistent with preeclampsia, after 20 WG.
Incidence of components of moderate and severe maternal morbidity | From inclusion up to discharge from hospital after delivery (max 30 days)
  Assessed during pregnancy and up to discharge from hospital after delivery (max 30 days)
  * Severe maternal morbidity (EPIMOMS composite criterion)
  * Postpartum hemorrhage (>500 mL), severe postpartum hemorrhage (>1000 mL), in the 24 hours of delivery as assessed by clinicians in charge of delivery
  * Cesarean delivery
  * Abruptio placenta
  * Maternal ICU admission
  * Maternal death
Incidence of components of moderate and severe perinatal morbidity | During pregnancy and up to discharge from hospital (max 30 days)
  * Perinatal death (stillbirth or neonatal death within 7 days of life)
  * Transfer to NICU
  * Miscarriage defined by fetal loss before 20 weeks of gestation
  * Stillbirth defined by intra uterine or perpartum fetal death at or after 20 WG
  * Perinatal death (stillbirth defined by intra uterine or peripartum fetal death at or after 20 WG or neonatal death within 7 days of life)
  * Gestational age at delivery
  * Prematurity < 37 WG, <34 WG, < 28WG
  * At delivery, Apgar score <7 at 5 min, umbilical cord pH <7.00 and Base excess >-12
  * Birth weight, birth weight percentile for gestational age, birth weight < 3° percentile for gestational age, birth weight < 10° percentile for gestational age
  * Transfer to NICU from delivery and up to discharge from hospital (max 30 days)
Impact of first-trimester PE screening on potential adverse events | From inclusion up to discharge from hospital (max 30 days)
  - Overmedicalization and iatrogenesis: total number of ultrasound exams during pregnancy, total number of prenatal visits (planned, emergency), total number of hospitalizations during pregnancy and number of days, antihypertensive treatment, heparin treatment
Aspirin side effects | From inclusion up to discharge from hospital (max 30 days)
  Aspirin side effects: epigastric pain during pregnancy, vaginal bleeding during pregnancy, other notable bleeding complication requiring hospitalization during pregnancy, nasal bleeding requiring packing during pregnancy, neonatal hemorrhage.
Women's anxiety 1 | At 20 WG (+/- 2 weeks) and day 2 postpartum (+/- 2 days)
  Anxiety will be assessed using the State-Trait Anxiety inventory State (STAI-S) self-administered questionnaire, validated in French, at 20 weeks of gestion (+/- 2 weeks) and at day 2 postpartum. All patients will be asked to complete self-administered questionnaires at 20 (+/2) WG and during the postpartum period (within 30 days after delivery) assessing women's satisfaction and women's anxiety. These questionnaires will be collected for women included until 31/01/2025."
Women's anxiety 2 | At 20 WG (+/- 2 weeks)
  Anxiety will be assessed using the self-administered Pregnancy-Related Anxiety Questionnaire (PRAQ-R2), validated in French, at 20 weeks of gestation (+/- 2 weeks). These questionnaires will be collected for women included until 31/01/2025.
Women's perception of information received and screening | At 20 WG (+/- 2 weeks)
  Assessed using self-administered questions developed for the trial at 20 weeks of gestation.
To evaluate the impact of first-trimester PE screening on costs and cost effectiveness 1 | From inclusion up to discharge from hospital (max 30 days)
  - Direct costs of prenatal, delivery, postnatal maternal care and neonatal care
To evaluate the impact of first-trimester PE screening on costs and cost effectiveness 2 | From inclusion up to discharge from hospital (max 30 days)
  - Total costs
To evaluate the impact of first-trimester PE screening on costs and cost effectiveness 3 | From inclusion up to discharge from hospital (max 30 days)
  - Incremental cost-effectiveness ratio: difference in costs/reduction in the incidence of severe perinatal morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Catherine DENEUX, MD, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (22):
- France (22):
  - CHU Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - Hôpital Femme Mère Enfant, Bron
  - Hôpital Antoine Béclère, Clamart
  - CHU Estaing, Clermont-Ferrand
  - Hôpital Intercommunal Créteil, Créteil
  - CHU Dijon Bourgogne, Dijon
  - CHU Lille, Lille
  - Hôpital de la conception et de la Timone, Marseille
  - Hôpital Nord, Marseille
  - CHRU de Nancy, Nancy
  - Hôpital Femme - Maternité, Nantes
  - Hôpital Armand Trousseau, Paris
  - Hôpital Cochin (site Port-Royal), Paris
  - Hôpital Saint-Joseph, Paris
  - CHI de Poissy, Poissy
  - Hôpital Sud Rennes, Rennes
  - CHU Charles Nicolle, Rouen
  - CHU Strasbourg, CMCO Schiltigheim, Strasbourg
  - Hôpital de Hautepierre, Strasbourg
  - Hôpital Paule de Viguier, Toulouse
  - Hôpital Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No